CLINICAL TRIAL: NCT05934916
Title: Early Application of Continuous Positive Airway Pressure in (Coronavirus Disease 2019) Patients at Risk of Obstructive Sleep Apnea
Brief Title: Early Application of Continuous Positive Airway Pressure in Coronavirus Patients at Risk of Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MS.21.07.1578.
Record Dates: First submitted 2023-06-24; First posted 2023-07-07 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2021-07

CONDITIONS: Covid19; Obstructive Sleep Apnea; CPAP Ventilation; Corona Virus Infection
Keywords: ( Coronavirus disease 2019); Coronavirus infections; sleep breathing disorder; obstructive sleep apnea
MeSH Terms: conditions — COVID-19; Sleep Apnea, Obstructive; Coronavirus Infections | interventions — Continuous Positive Airway Pressure; Oxygen Inhalation Therapy

STUDY DESIGN:
Intervention Model Description: Non-CPAP group will receive medical treatment plus oxygen therapy according to recommendation of protocol of the Egyptian Ministry of Health 2020 and CPAP group as in Non-CPAP group plus using CPAP.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous Positive Airway Pressure (CPAP) group in (Coronavirus disease 2019) patients (Experimental): receive medical treatment plus oxygen therapy according to recommendation of protocol of the Egyptian Ministry of Health 2020 and using Continuous Positive Airway Pressure (CPAP)
  Interventions: Device: CPAP ( Continuous positive airway pressure); Device: oxygen therapy
- Non-CPAP group (Experimental): Non-CPAP group will receive medical treatment plus oxygen therapy according to recommendation of protocol of the Egyptian Ministry of Health 2020
  Interventions: Device: oxygen therapy

INTERVENTIONS:
Device: CPAP ( Continuous positive airway pressure) — The enrolled eighty patients were simply randomized into two equal groups: Non-CPAP group and CPAP group using a computer-generated table of random numbers. The group allocation was concealed in sequentially numbered, sealed, and opaque envelopes. Patients were selected from isolation center in Mansoura University hospital,Non-CPAP group will receive medical treatment plus oxygen therapy according to recommendation of protocol of the Egyptian Ministry of Health 2020 and CPAP group as in Non-CPAP group plus using CPAP.
  Arms: Continuous Positive Airway Pressure (CPAP) group in (Coronavirus disease 2019) patients
Device: oxygen therapy — both groups will receive oxygen

SUMMARY:
This was an experimental clinical trial, Aim: To evaluate the role of early use of Continuous Positive Airway Pressure (CPAP) in management of moderate to severe Coronavirus disease 2019 patients at risk of Obstructive Sleep Apnea, enrolled patients are randomized into two equal groups;Non- CPAP group and CPAP group. Non-CPAP group will receive medical treatment plus oxygen therapy according to recommendation of protocol of the Egyptian Ministry of Health 2020 and CPAP group as in Non-CPAP group plus using CPAP.

DETAILED DESCRIPTION:
steps included

1. Clinical Assessment:

   Full history taking were taken from the enrolled Coronavirus disease 2019patients including age, occupation, medical history and special habits), Coronavirus disease 2019 symptoms (e.g., fever, dyspnea, fatigue, loss of smell or taste, (gastrointestinal tract) symptoms….) as well as all obstructive sleep apnea symptoms (e.g., Snoring, Insomnia, Excessive day time sleepiness, witnessed apnea, …).
2. II. Scales & Questionnaires:

   * Epworth Sleepiness Scale (ESS) It's designed to assess the degree of daytime sleepiness.
   * - Berlin Questionnaire
   * - (Snoring, Tiredness, observed apnea, high blood pressure, body mass Index, age, neck circumference and male Gender questionnaire: This scoring system composed of 8 items that are graded from 0 to 8 according to Yes/No responses (score: 1/0).
3. III. Radiological investigations
4. IV. Laboratory Investigations Blood gases, complete blood picture, etc
5. . CPAP application Auto-CPAP with continuous nocturnal administration or at least4- 6hours /night and during day naps, for more than 70% of nights from the first night of admission to isolation center

ELIGIBILITY:
Inclusion Criteria:

* patients age above 18 years, diagnosed with moderate to severe (Coronavirus disease 2019) and at risk of Obstructive Sleep Apnea as well as confirmed nasopharyngeal swab positive for (Severe acute respiratory syndrome coronavirus 2) ( by (polymerase chain reaction).

Exclusion Criteria:

* patients were excluded from the study if their age <18 years, hypercapnic, unstable cardiorespiratory (shock) status or respiratory arrest and if there are any contraindications for ( Continuous Positive Airway Pressure (CPAP) mask use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Survival n (%), In hospital mortality , Duration of hospital stay, Need for invasive ventilation | 8 months

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University, Al Mansurah, Al Dakahlia, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol